CLINICAL TRIAL: NCT04261920
Title: Study on Efficacy and Safety of Huangqi Guizhi Wuwu Decoction Treatment for Oxaliplatin Induced Peripheral Neurotoxicity: a Protocol for a Randomized, Controlled, Double-blind, Multi-center Trial
Brief Title: Clinical Trial Scheme of Huangqi Guizhi Wuwu Decoction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FM-P8-2018060101
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Oncology
Keywords: Oxaliplatin induced peripheral neurotoxicity; Clinical curative effect
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with colorectal cancer diagnosed by histopathological examination; patients after radical resection of colorectal cancer confirmed by histopathological examination, staged as high-risk II stage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single decoction group: Huangqi Guizhi Wuwu decoction (Experimental): The dosage of granules: Sheng huangqi granule 5.5g/bag, Guizhi granule 0.9g/bag, Baishao granule 1.6g/bag, Ganjiang granule 1.7g/bag, Dazao granule 7g/bag. Take twice a day, infused with warm water. Consistently used during patients receiving XELOX5 adjuvant chemotherapy for at least 12 weeks (every 3 week is a cycle, 4 cycles)
  Interventions: Drug: Huangqi Guizhi Wuwu decoction
- Simulator group: Huangqi Guizhi Wuwu decoction Placebo (Placebo Comparator): The control group took placebo twice a day, infused with warm water. Consistently used during patients receiving XELOX5 adjuvant chemotherapy for at least 12 weeks (every 3 week is a cycle, 4 cycles)
  Interventions: Drug: Huangqi Guizhi Wuwu decoction

INTERVENTIONS:
Drug: Huangqi Guizhi Wuwu decoction — The experimental group took Huangqi Guizhi Wuwu decoction twice a day, infused with warm water. Consistently used during patients receiving XELOX5 adjuvant chemotherapy for at least 12 weeks (every 3 week is a cycle, 4 cycles).
  The control group took placebo twice a day, infused with warm water. Consistently used during patients receiving XELOX5 adjuvant chemotherapy for at least 12 weeks (every 3 week is a cycle, 4 cycles).
  Other Names: Huangqi Guizhi Wuwu decoction placebo

SUMMARY:
To evaluate the efficacy and safety of Huangqi Guizhi Wuwu decoction in preventing oxaliplatin induced peripheral neurotoxicity.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate whether the preventive effect of Huangqi Guizhi Wuwu decoction on oxaliplatin induced peripheral neurotoxicity is better than that of simulator, and to provide evidence-based medicine basis for the clinical promotion of single medicine granule. This trial purpose is to evaluate the efficacy and safety of Huangqi Guizhi Wuwu decoction in preventing oxaliplatin induced peripheral neurotoxicity. This trial design type is a randomized, controlled, double-blind, multicenter clinical study was conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with colorectal cancer diagnosed by histopathological examination; patients after radical resection of colorectal cancer confirmed by histopathological examination, staged as high-risk II stage (according to CSCO guidelines for diagnosis and treatment of colorectal cancer) or III stage, IV stage (metastatic lesions have been radical resection); 2. Patients who are suitable for receiving oxaliplatin plus capecitabine regimen as adjuvant chemotherapy for 6 months, the cumulative dose of oxaliplatin are expected to exceed 520mg/m2 at least; 3. Aged from 18 to 75 years old, males or females; 4. ECOG score ranges from 0 to 1 5. Seven days before treatment, the functions of major organs (heart, liver, kidney, bone marrow) meet the following criteria:

1. Standard of blood routine examination (without blood transfusion within 14 days) i. Hemoglobin (HB) ≥90g/L； ii. Absolute Neutrophil Count(ANC) ≥1.5×109/L；. iii. Platelet (PLT) ≥80×109/L.
2. Biochemical examination should meet the following standards:

   * Total bilirubin(TBIL) ≤1.5 times upper normal limit(ULN);

     * Alanine aminotransferase(ALT) and Aspartate aminotransferase(AST) ≤2.5 times ULN；

       ③Serum creatinine （Cr）≤1.5 times ULN or Creatinine clearance(CCr) ≥60ml/min; 6.Expected survival time≥12 months; 7. For subjects who have used other chemotherapeutic drugs in the past, they need to go through a clearance period of at least 4 weeks before entering this trial.

       8. The patient who will sign the informed consent form

Exclusion Criteria:

1. Patients with original nervous system diseases, including peripheral neuropathy and central neuropathy;
2. Those who are allergic to oxaliplatin or the ingredients of this traditional Chinese medicine;
3. Clinical symptoms of patients with severe damp-heat syndrome of colorectal cancer include: dry mouth, bitter taste in the mouth, sticky sensation in mouth, yellow urine, dry stool, red tongue with yellow ,thick and greasy fur;
4. Patients with neurological disease caused by electrolyte disorders or diabetes;
5. Patients with symptoms of nerve compression caused by various causes;
6. At the same time, patients who receive other neuroprotective therapy, including nerve growth factor, vitamin B and calcium-magnesium mixture;
7. Patients who were treated with oxaliplatin for chemotherapy before;
8. Patients who need radiotherapy within half a year after operation;
9. Pregnant or lactation period women;
10. Patients with cognitive impairment or psychosis;
11. Other patients the investigator considers unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-01-03 (Actual); Primary Completion 2023-01-02 (Estimated); Study Completion 2023-03-02 (Estimated)

PRIMARY OUTCOMES:
incidence of chronic neurotoxicity | 3 years
  Differences in the incidence of chronic neurotoxicity of grade 2 and above during and after treatment

SECONDARY OUTCOMES:
incidence of acute neurotoxicity | 3 years
  Difference in the incidence of acute neurotoxicity
Time of occurrence of chronic toxicity | 3 years
  Time of occurrence of chronic toxicity to grade 2 and 3
main symptoms | 3 years
  Incidence and severity of main symptoms
Recovery time of neurotoxicity | 3 years
  Recovery time of grade 2 and 3 neurotoxicity
Cumulative dose of oxaliplatin and the proportion of patients | 3 years
  Cumulative dose of oxaliplatin and the proportion of patients who stop using oxaliplatin because of neurotoxicity
myelosuppression | 3 years
  Incidence of myelosuppression
nausea, vomiting, diarrhea, and hand-foot syndrome | 3 years
  Incidence of nausea, vomiting, diarrhea, and hand-foot syndrome

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Hospital of Nanjing University of TCM, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wei XM, Chen XF, Shu P, Jiang ZW, Wu XY, Zou X, Chen K, Shen B, Hu WW, Lu W, Shen WX, Li L, Wang JY, Zhao FJ, Yin QF, Cheng HB, Gu YH. Study on efficacy and safety of Huangqi Guizhi Wuwu decoction treatment for oxaliplatin induced peripheral neurotoxicity: A protocol for a randomized, controlled, double-blind, multicenter trial. Medicine (Baltimore). 2020 May 29;99(22):e19923. doi: 10.1097/MD.0000000000019923. PMID 32481364